CLINICAL TRIAL: NCT01286688
Title: Randomized, 2-way Crossover Bioequivalence Study of Terbinafine Hydrochloride Tablets, 250 mg and Lamisil® 250 mg Tablets in Healthy Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Terbinafine Hydrochloride Tablets, 250 mg of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Dr. Ramakrishna Bangaru/Assistant Manager, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01361
Record Dates: First submitted 2011-01-26; First posted 2011-01-31 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Fasting
Keywords: Bioequivalence; crossover; Terbinafine hydrochloride; Fasting
MeSH Terms: conditions — Fasting | interventions — Terbinafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Terbinafine Hydrochloride (Experimental): Terbinafine Hydrochloride Tablets, 250 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Terbinafine Hydrochloride Tablets, 250 mg
- Lamisil® 250 mg Tablets (Active Comparator): Lamisil® 250 mg Tablets of Novartis
  Interventions: Drug: Terbinafine Hydrochloride Tablets, 250 mg

INTERVENTIONS:
Drug: Terbinafine Hydrochloride Tablets, 250 mg — Terbinafine Hydrochloride Tablets, 250 mg of Dr. Reddy's Laboratories Limited.
  Other Names: Lamisil® 250 mg Tablets

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of terbinafine hydrochloride 250 mg tablets versus Lamisil® 250 mg tablets administered as 1 x 250 mg tablet under fasting conditions.

DETAILED DESCRIPTION:
Randomized, 2-way crossover, bioequivalence study of Terbinafine hydrochloride 250 mg tablets and Lamisil® 250 mg Tablets administered as 1 x 250 mg tablet in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may be done using different media (e.g. radio, newspaper, Anapharm Web site, Anapharm volunteers' data base). ---Subjects must meet all of the following criteria in order to be included in the study:
* Subjects will be females and/or males, smokers and/or non-smokers, 18 years of age and older.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical sub-investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90 mm Hg; or heart rate less than 50 bpm) at screening.

Subjects with BMI ≥ 30.0.

* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical sub-investigator, contraindicates the subjects participation in this study.
* History of allergic reactions to terbinafine hydrochloride or other related drugs (e.g.naftifine).
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin;examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin,ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine), use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural products, vitamins, garlic as supplement)within 7 days prior to administration of study medication, except for topical products without systemic absorption or oral contraceptives.
* Subjects who have a depot injection or an implant of any drug (except for depot injection or implant used as method of contraception) 3 months prior to administration of study medication.
* Subjects with a history of any previous liver disease.

Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follow:

* less than 300 mL of whole blood within 30 days or
* 300 mL to 500 mL of whole blood within 45 days or
* more than 500 mL of whole blood within 56 days. •Smoking more than 25 cigarettes per day.

Additional exclusion criteria for females only:

* Breast-feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).
* Female subjects of childbearing potential who have had unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. The acceptable methods of contraception are:

  * Condom + spermicide
  * Diaphragm + spermicide
  * Intrauterine contraceptive device (placed at least 4 weeks prior to study drug administration)
  * oral contraceptives (starting at least 4 weeks prior to study drug administration)
  * Implant (e.g. Norplant®) (starting at least 4 weeks prior to study drug administration)
  * Depot injection of a progestogen drug (e.g. Depo-Provera®) (starting at least 4 weeks prior to study drug administration)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2002-01; Primary Completion 2002-02 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence study based on Cmax parameter | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bicrell, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Québec, Canada